CLINICAL TRIAL: NCT05132543
Title: Studying Human Cognition and Neurological Disorders Using ÂµECoG Electrodes
Brief Title: Neural Basis of Cognition
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00072892; 5R01DC019498 (NIH)
Record Dates: First submitted 2021-10-25; First posted 2021-11-24 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wireless µECoG Prosthesis for Speech (Experimental)
  Interventions: Device: High density micro-electrocorticography for neural speech prothesis

INTERVENTIONS:
Device: High density micro-electrocorticography for neural speech prothesis — ECoG electrodes are thin, high-density, flexible electrode arrays used for recording electrophysiological signals from the brain.

SUMMARY:
The overall purpose of this study is to better understand human cognition and human epilepsy by working with patients undergoing clinical treatment for pharmacologically resistant epilepsy. The investigators will investigate human cognition by conducting controlled experiments that focus on sensory, motor, and cognitive phenomena such as sensory processing, memory, and language. The investigators will also examine the neural underpinnings of epilepsy during both sleep and wakefulness to better understand both the foundations of epilepsy and how epilepsy affects cognition. The investigators hope to use these data to have a better understanding of cognition, epilepsy, and how the two interact. This will potentially lead to better markers for seizure onsets as well as epilepsy more generally. For this research, the investigators will use μECoG arrays manufactured by commercial partners. These arrays have passed all major ISO 10993 bio-compatibility tests. Based on this characterization and use in the intraoperative setting (limited duration and supervised usage), these devices pose a minimal risk to participants. Data will be analyzed and protected using the Duke SSRI protected research data network.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects will come from adult and pediatric patients (between the ages of 12 and 18) undergoing surgery for the treatment of pharmacologically resistant epilepsy, brain tumor resection, brain mass resection, or deep brain stimulation (DBS) for the first time
* Proficient English speakers
* No Major cognitive impairment

Exclusion Criteria:

* Previous DBS procedure
* Subject unable to consent to study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-09-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Evoked signal-to-noise analysis human brain. | Intraoperative data collection period, 20 minutes
  This study will compare the neural response sensitivity of intraoperative µECoG recording to those of in-unit recordings with macro-ECoG and SEEG. The strength and reliability of the high gamma (HG) response are critical for speech decoding algorithms. For all recordings, the HG power modulation ratio over baseline during speech perception and production will be measured and compared with non-parametric statistical tests.
Percentage of phoneme decoding accuracy as measured by linear decoding model | Intraoperative data collection period, 20 minutes
Number of HG power modulation as measured by signal power. | Intraoperative data collection period, 20 minutes
Number of kriging resolution as measured by signal power. | Intraoperative data collection period, 20 minutes

SECONDARY OUTCOMES:
Number of serious adverse events as measured by medical record review | Implantation to Three-months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Gregory B Cogan, PhD, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: Yes
Following completion of this project and 8 months after acceptance of the primary manuscript(s), the research data will be made available to the scientific community through public repository for neurophysiological data (e.g. Pennsieve and crcns.org) for both research and educational purposes. Recordings from clinical and research electrodes will be de-identified.
  The investigators will also include the relevant task data, electrode coordinates in MNI and subject specific space, essential de-identified clinical data using NINDS Common Data Elements (age, sex, duration of epilepsy, epilepsy etiology, preoperative imaging findings), schematics of seizure-onset areas, and any relevant scripts needed to manipulate the data. All data will be reviewed prior to upload to ensure they contain no PHI and will be stripped of voice recordings and be HIPAA compliant.
Supporting Information: ICF, Analytic Code
Time Frame: Following completion of this project and 8 months after acceptance of the primary manuscript(s), the research data will be made available to the scientific community.
Access Criteria: DANDI repository